CLINICAL TRIAL: NCT04258293
Title: Diabetes Screening in Patients on Long-Term Glucocorticoid Therapy
Acronym: DIACORT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOUILLET 2018-2
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Glucocorticosteroid; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients on prolonged corticosteroid therapy (more than three months)
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — fasting venous glycemia, venous glycemia after sugar loading, glycated hemoglobin and platelet count

SUMMARY:
Glucocorticoids are widely prescribed in the treatment of many inflammatory, autoimmune or allergic diseases, but also in transplant patients or patients with malignant hematological diseases (leukaemia, lymphoma, myeloma, etc.). They have many side effects, including effects on carbohydrate metabolism.

Corticosteroids are diabetogenic because they disrupt pancreatic insulin secretion and decrease the insulin sensitivity of target tissues (liver, muscle, adipose tissue).

The use of glucocorticoids may lead to the development of corticosteroid-induced diabetes in non-diabetic patients.

Corticosteroid-induced diabetes is frequently found in clinical practice. Incidence figures for corticosteroid-induced diabetes vary widely.

Case-control studies show odds ratios of corticosteroid-induced diabetes onset ranging from 1.36 and 2.23. In two of these studies, the diagnostic criterion was the prescription of a hypoglycemic treatment. Smaller studies, retrospective or prospective, show incidence rates of corticosteroid-induced diabetes ranging from 8.8 to 52%. This difference in incidence rates is explained by the different glucocorticoid doses, glucocorticoid durations, conditions requiring glucocorticoid therapy, and diagnostic criteria for corticosteroid-induced diabetes that vary from study to study. In kidney transplantation, diabetes concerns 16% of patients before the age of 40, and up to 52% after the age of 50. The diagnostic criteria used in the literature are often fasting and post prandial glycemia. The differences in incidence rates found with these two diagnostic methods can be explained by the pharmacokinetics of glucocorticoids. The main glucocorticoids prescribed have a duration of action of 12 to 16 hours. As they are generally prescribed in the morning as a single daily dose, fasting morning blood glucose levels are often normal while postprandial blood glucose levels are increased. This observation has been presented in 2 studies. However, the 2 diagnostic criteria were not statistically compared in these studies.

While according to the American Diabetes Association, the 3 criteria used to diagnose diabetes are fasting glycemia, glycemia 2 hours after an oral glucose load of 75 g and glycated hemoglobin, these last 2 diagnostic criteria are, to the investigator's knowledge, not used in the scientific literature to screen for corticosteroid-induced diabetes.

In current practice, the diagnostic criteria used are disparate. To date, there are no studies that have determined which diagnostic criterion is the most effective in screening for corticosteroid-induced diabetes. The current recommendations recommend early diagnosis and treatment in order to achieve satisfactory glycemic control as quickly as possible. These recommendations have been shown to be effective in reducing the risk of degenerative complications of diabetes, but it is important to screen for corticosteroid-induced diabetes with the most relevant diagnostic criterion in order to optimise its management.

ELIGIBILITY:
Inclusion Criteria:

* Person who has orally provided voluntary informed consent.
* Patient with an indication for prolonged corticosteroid therapy (more than three months)
* Non-diabetic patient

Exclusion Criteria:

* Person not affiliated to or not benefiting from national health insurance system
* Person subject to legal protection (guardianship, curatorship)
* Pregnant or breastfeeding woman
* Adult unable to provide consent
* Minor
* Evidence of fasting venous blood glucose greater than 1.26 g/L, or Glycated haemoglobin greater than 6.5% at the time of initial blood sampling before glucocorticoid treatment.
* Patient who had received corticosteroid therapy within 3 months prior to the study
* Patient with hemoglobin less than 10 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatients and outpatients
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
fasting venous glycemia | an average of 3 months
venous glycemia after sugar loading | an average of 3 months
Glycated Hemoglobin | an average of 3 months
Platelet Count | an average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France